CLINICAL TRIAL: NCT05571501
Title: Measuring Normal and Impaired Walking in Children Using the GAITRite Walkway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: GOSHCC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10NS14; 11/LO/1889 (Other: NRES)
Record Dates: First submitted 2015-04-23; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Typically Developing Children; Talipes Equino Varus; Paediatric Orthopaedic; Paediatric Neurological

STUDY DESIGN:
Intervention Model Description: The tool used for this study has been and was used for routine patient care, but was a novel diagnostic assessment for the typically developing (norms) and some of the clinical groups included. The clinical groups were compared to norms, both had the same diagnostic assessment so there was no control group who did not have the assessment
Masking Description: All children recruited underwent the GAITRite assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typically developing children (Active Comparator): 500 children aged 1-18 male and female will be recruited from local schools, after school clubs and playgroups.
  Each child will complete a screening form following appropriate information and consent process. Each child will then complete the walking assessment which takes 15 minutes in total
  Interventions: Device: Gait assessment using the GAITRIte walkway
- Clinical groups (Active Comparator): Children will be recruited through their patient journey. Families who consent to participation will complete the screening form and the GAITRite walking assessment as part of their pre-planned clinical followup in outpatient clinics.
  One group of children will be assessed at one time point, whilst a second group of children with progressive orthopaedic conditions or treatment will be assessed at intervals to give longitudinal data
  Interventions: Device: Gait assessment using the GAITRIte walkway

INTERVENTIONS:
Device: Gait assessment using the GAITRIte walkway — 10-20 walking assessment using the GAITRite walkway
  Other Names: GAITRite

SUMMARY:
Walking measurement in children is important but there are challenges associated with obtaining reliable repeatable data in a clinical setting that is meaningful and easy to interpret. This study set out to develop a new way to collect, record, and interpret walking data that is suitable for the clinical environment. Developmental percentile charts were selected as they are widely recognised and easily interpreted.

DETAILED DESCRIPTION:
The primary output of the main cohort of typically developing children is the developmental percentile charts.

These will be then used to present the clinical longitudinal data against a normal backdrop of developmental changes in children.

This has multiple clinical applications in many of the children assessed by physiotherapy at GOSH and more widely Nationally and internationally

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 100m

Exclusion Criteria:

* recent fracture or musculoskeletal injury which would affect gait

Ages: 10 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 702 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Gait data recorded via GAITRite software | For the duration of the study measured once for typically developing and at multiple clinic visits over 24 months for clinical groups
  Continuous numeric data summarising walking performance and characteristics

SECONDARY OUTCOMES:
demographic and clinical outcome data | 30 to 60 mins to collect relevant data at a single time point, with an update to include additional admissions over 24months
  surgical history (where relevant)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Alderson, PhD, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only summary centile charts for norms will be available with no individual identifiers

REFERENCES:
- [Background] Wood M, Cleary MA, Alderson L, Vellodi A. Changes in gait pattern as assessed by the GAITRite walkway system in MPS II patients undergoing enzyme replacement therapy. J Inherit Metab Dis. 2009 Dec;32 Suppl 1:S127-35. doi: 10.1007/s10545-009-1103-2. Epub 2009 Mar 25. PMID 19319660
- [Background] Bladen M, Alderson L, Khair K, Liesner R, Green J, Main E. Can early subclinical gait changes in children with haemophilia be identified using the GAITRite walkway. Haemophilia. 2007 Sep;13(5):542-7. doi: 10.1111/j.1365-2516.2007.01429.x. PMID 17880441
- [Result] Alderson LM, Joksaite SX, Kemp J, Main E, Watson T, Platt FM, Cortina-Borja M. Age-related gait standards for healthy children and young people: the GOS-ICH paediatric gait centiles. Arch Dis Child. 2019 Aug;104(8):755-760. doi: 10.1136/archdischild-2018-316311. Epub 2019 Mar 25. PMID 30910816